CLINICAL TRIAL: NCT02015416
Title: A Phase 1 Open Label, Multicenter, Multiple Ascending Dose Trial Evaluating the Safety, Tolerability and Immunogenicity of Intramuscular Recombinant NY-ESO-1 Protein With GLA-SE Adjuvant in Patients With Unresectable or Metastatic Cancer
Brief Title: A Phase 1 Trial of NY-ESO-1 With GLA-SE in Patients With Unresectable or Metastatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Immune Design, a subsidiary of Merck & Co., Inc. (Rahway, New Jersey USA) (Industry)
Responsible Party: Sponsor
Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IDC-G305-2013-001
Record Dates: First submitted 2013-12-13; First posted 2013-12-19 (Estimated); Last update posted 2017-08-17 (Actual); Status verified 2017-08

CONDITIONS: Melanoma; Ovarian Cancer; Sarcoma; Non-small Cell Lung Cancer; Breast Cancer
Keywords: Melanoma; Ovarian cancer; Sarcoma; Non-small cell lung cancer; NSCLC; Breast cancer
MeSH Terms: conditions — Melanoma; Ovarian Neoplasms; Sarcoma; Carcinoma, Non-Small-Cell Lung; Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: Phase 1, open label, multicenter ascending dose study.
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- IDC-G305 (Experimental): NY-ESO-1 recombinant protein together with GLA-SE
  Interventions: Biological: IDC-G305

INTERVENTIONS:
Biological: IDC-G305 — NY-ESO-1 recombinant protein together with GLA-SE

SUMMARY:
This is a Phase I, multi-center, multiple ascending dose study to evaluate the clinical safety and immune response of IDC-G305 when injected intramuscularly in patients with unresectable or metastatic cancer. IDC-G305 is an immunotherapy consisting of recombinant NY-ESO-1 antigen and the adjuvant, GLA-SE. The goal is for IDC-G305 to stimulate the body's immune system to fight the spread and growth of cancer for patients whose tumors include the NY-ESO-1 protein. Patients with melanoma, ovarian, renal cell or non-small cell lung cancer may be considered for the trial.

DETAILED DESCRIPTION:
This is a Phase 1, open label, multicenter, multiple ascending dose trial of IDC-G305 administered by intramuscular injection in a 3+3 sequential dose escalation design. IDC-G305 is an immunotherapy consisting of recombinant NY-ESO-1 antigen and the adjuvant, GLA-SE. Patients with unresectable, relapsed or metastatic cancer but with low disease burden and indolent disease course may be considered for the trial. Tumors must express the NY-ESO-1 gene signature and tumor types that will be studied are: melanoma, ovarian, sarcoma,non-small cell lung and breast cancer.

Each of three dose level cohorts will be treated contingent upon absence of dose limiting toxicity (DLT) and acceptable safety data for the preceding cohort. Initially, three patients will be scheduled to receive IDC-G305 in each dose level cohort. Dose escalation will be contingent upon the assessment of safety data obtained during the initial injections.

Patients will be evaluated at baseline and at regular intervals for safety and immune response. Both cellular and humoral immunogenicity will be explored.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of melanoma, ovarian cancer, sarcoma, breast cancer or non-small cell lung cancer (NSCLC)
* Unresectable, relapsed and/or metastatic cancer with minimal or low disease burden. Disease may or may not be measurable and should not be rapidly progressive. Inadequate response, relapse and/or unacceptable toxicity with one or more prior systemic, surgical, or radiation cancer therapies, except patients with NSCLC and breast cancer who must have experienced an inadequate response and/or unacceptable toxicity with two or more prior systemic, surgical, or radiation cancer therapies.
* Cancer expresses NY-ESO-1
* ≥ 18 years of age
* Life expectancy of ≥ 6 months
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* ECG without evidence of clinically significant arrhythmia or ischemia
* Negative pregnancy test for females of childbearing potential

Exclusion Criteria:

* Pregnant or nursing
* Vaccine or other therapy directed against NY-ESO-1 at any time in the past and any investigational therapy within three weeks prior to IDC-G305 dosing
* Significant immunosuppression
* Cancer chemotherapy, G-CSF or GM-CSF within three weeks prior to the first study treatment
* Significant autoimmune disease
* Myocardial infarction within six months of treatment, active cardiac ischemia or Grade III or IV heart failure
* Inadequate hematology or chemistry profiles
* History of other cancer within three years
* Active, concurrent or recent infection, including tuberculosis, hepatitis B, hepatitis C or HIV
* Uveal melanoma
* Brain metastases considered unstable

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability | Up to 1 year after last vaccination
  To evaluate the safety and tolerability of multiple ascending doses of intramuscular (IM) IDC-G305

SECONDARY OUTCOMES:
Immunogenicity | Approximately 12 weeks
  The secondary objective is to evaluate the humoral and cellular immunogenicity of multiple ascending doses of intramuscularly administered IDC-G305

CONTACTS AND LOCATIONS:
Overall Officials: Kunle Odunsi, MD PhD, Principal Investigator — Roswell Park Cancer Institute
Locations (4):
- United States (4):
  - Scottsdale Healthcare, Scottsdale, Arizona
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Karmanos Cancer Institute, Detroit, Michigan
  - Roswell Park Cancer Institute, Buffalo, New York

IPD SHARING:
Plan to Share IPD: No